CLINICAL TRIAL: NCT01766661
Title: Prospective Multicenter Randomized Controlled Trial Comparing Postoperative Complications and Quality of Life in Low Rectal Cancer Surgery Between Coloanal Anastomosis and Lateral Ileostomy Versus Two-Stage Turnbull-Cutait Coloanal Anastomosis
Brief Title: Prospective Multicenter Randomized Controlled Trial On Two-Stage Turnbull-Cutait Coloanal Anastomosis For Rectal
Acronym: TURNBULL-BCN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Sebastiano Biondo, PhD, MD, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TURNBULL-BCN-01; PR174/11 (Other: CEIC Hospital Universitari de Bellvitge)
Record Dates: First submitted 2013-01-10; First posted 2013-01-11 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Rectal Neoplasm
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coloanal anastomosis with ileostomy (Active Comparator): Hand-sewn coloanal anastomosis protected by a loop ileostomy
  Interventions: Procedure: Hand-sewn coloanal anastomosis; Procedure: Ultralow anterior rectal resection with total mesorectal excision
- Two stage Turnbull-Cutait anastomosis (Experimental): Two staged coloanal anastomosis without protective ileostomy (Turnbull-Cutait procedure).
  Interventions: Procedure: Two staged Turnbull-Cutait procedure; Procedure: Ultralow anterior rectal resection with total mesorectal excision

INTERVENTIONS:
Procedure: Hand-sewn coloanal anastomosis — After low anterior rectal resection due to low rectal neoplasm patients undergo intestinal reconstructions as hand-sewn coloanal anastomosis with protective loop ileostomy.
  Arms: Coloanal anastomosis with ileostomy
Procedure: Two staged Turnbull-Cutait procedure — After low anterior rectal resection due to low rectal neoplasm patients undergo intestinal reconstructions as two staged Turnbull-Cutait procedure anastomosis without protective ileostomy.
  Arms: Two stage Turnbull-Cutait anastomosis
Procedure: Ultralow anterior rectal resection with total mesorectal excision — Standard ultralow anterior rectal resection with total mesorectal excision

SUMMARY:
The aim of this study is to decrease the morbidity by 30% using the Turnbull-Cutait procedure in comparison to the standard surgery for low rectal cancer. The investigators compare quality of life, faecal incontinence and recurrence of neoplasm in patients who received standard colo-anal anastomosis with protective ileostomy or two-staged Turnbull-Cutait colo-anal anastomosis after Low Anterior Resection for rectal cancer.

DETAILED DESCRIPTION:
Anastomotic leak represents the most frequent complication after rectal cancer surgery and a lateral covering ileostomy is usually performed to reduce its incidence. Other important consequences of rectal cancer surgery are alterations in bowel habits and function and a negative impact on quality of life. This prospective, randomized, multicenter and controlled trial compares post-operative complications, quality of life, faecal incontinence and recurrence rate in patients treated for low rectal cancer with colo-anal anastomosis protected by a lateral ileostomy or with a two-staged Turnbull-Cutait colo-anal anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with adenocarcinoma of the lower-middle third of the rectum proctoscopy established by rigid proctoscopy, with histological confirmation and candidates of colo-anal anastomosis;
* Patients over 18 years and under 75 years, who can tolerate neoadjuvant and surgical treatment;
* Patients who undergo an ultra-low anterior rectal resection with total mesorectal excision and nerve and sphincter-sparing with curative intention
* Any extension of the primary tumor (T 1-2-3-4) according to the TNM classification;
* Patients with or without lymph node metastasis (N - / +) and with or without resectable distant metastases;
* Patients clinically without fecal incontinence prior to the current illness and with a Wexner incontinence Score less than or equal to 5;
* Patients ASA I, II or III and adequate hematological, renal and hepatic function;
* Patients who signed informed consent.

Exclusion Criteria:

* Altered cognitive state(eg mental retardation or dementia) that prevents collaboration in the study or patients who can neither read nor write
* Fecal incontinence (Wexner equal to or greater than 6);
* Previous surgery or proctological, colonic and anorectal functional disease
* Diagnosis of synchronous colorectal or any other active neoplasm;
* Patients ASA IV, V;
* Pregnancy and lactation;
* Rejection of the patient to sign the consent form.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-01; Primary Completion 2019-03 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
post-operative morbidity | within the first 30 days after surgery

SECONDARY OUTCOMES:
Quality of life | 3 years
  by COREFO questionnaire.
Fecal incontinence | 3 years
  by Wexner Incontinence Score
local and/or distant recurrence of neoplasm | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Sebastiano Biondo, MD, Phd, Principal Investigator — Bellvitge University Hospital
Locations (4):
- Istituto Nazionale Tumori "Fondazione G, Pascale" - IRCCS, Naples, Italy
- Spain (3):
  - Corporació Sanitària Parc Taulí Hospital Universitari, Sabadell, Barcelona
  - Vall d'Hebron Universitary Hospital, Barcelona
  - Bellvitge University Hospital, Barcelona

REFERENCES:
- [Derived] Biondo S, Barrios O, Trenti L, Espin E, Bianco F, Falato A, De Franciscis S, Solis A, Kreisler E; TURNBULL-BCN Study Group. Long-Term Results of 2-Stage Turnbull-Cutait Pull-Through Coloanal Anastomosis for Low Rectal Cancer: A Randomized Clinical Trial. JAMA Surg. 2024 Sep 1;159(9):990-996. doi: 10.1001/jamasurg.2024.2262. PMID 38985480
- [Derived] Biondo S, Trenti L, Espin E, Bianco F, Barrios O, Falato A, De Franciscis S, Solis A, Kreisler E; TURNBULL-BCN Study Group. Two-Stage Turnbull-Cutait Pull-Through Coloanal Anastomosis for Low Rectal Cancer: A Randomized Clinical Trial. JAMA Surg. 2020 Aug 1;155(8):e201625. doi: 10.1001/jamasurg.2020.1625. Epub 2020 Aug 19. PMID 32492131
- [Derived] Biondo S, Trenti L, Galvez A, Espin-Basany E, Bianco F, Romano G, Kreisler E; Turnbull-BCN study group. Two-stage Turnbull-Cutait pull-through coloanal anastomosis versus coloanal anastomosis with protective loop ileostomy for low rectal cancer. Protocol for a randomized controlled trial (Turnbull-BCN). Int J Colorectal Dis. 2017 Sep;32(9):1357-1362. doi: 10.1007/s00384-017-2842-4. Epub 2017 Jun 30. PMID 28667499